CLINICAL TRIAL: NCT06719700
Title: A Prospective Phase II Study of Concurrent Chemoradiotherapy Combined With Toripalimab and Surufatinib in the Treatment of Limited-Stage Small Cell Lung Cancer
Brief Title: Concurrent Chemoradiotherapy Combined With Toripalimab and Surufatinib in the Treatment of Limited-Stage Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-10123
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Toripalimab; Surufatinib; Chemoradiotherapy; Limited-stage Small Cell Lung Cancer (LS-SCLC)
Keywords: Toripalimab; Surufatinib; Chemoradiotherapy; Limited-stage small cell lung cancer (LS-SCLC); Immunotherapy consolidation
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Drug Therapy; Immunotherapy; Radiotherapy; toripalimab; surufatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The study group (Experimental): In this single-arm, patients are planned to receive four cycles of etoposide combined with either cisplatin or carboplatin, along with toripalimab and surufatinib. During chemotherapy, patients will undergo concurrent radiotherapy. Following chemoradiotherapy, consolidation treatment with toripalimab and surufatinib will be administered. Prophylactic cranial irradiation (PCI) is recommended prior to the initiation of immunotherapy consolidation.
  Interventions: Drug: Chemotherapy; Drug: Immunotherapy; Drug: Angio-immuno kinase inhibitor; Radiation: radiotherapy; Radiation: Prophylactic Cranial Irradiation; Drug: Consolidation Therapy with Toripalimab and Surufatinib

INTERVENTIONS:
Drug: Chemotherapy — Etoposide combined with cisplatin or carboplatin, administered every three weeks for a total of four cycles.
Drug: Immunotherapy — Toripalimab was administered concurrently with chemotherapy, every three weeks for four cycles.
Drug: Angio-immuno kinase inhibitor — Oral surufatinib 200 mg once daily (q.d.), given on days 1-14 of each chemotherapy cycle.
Radiation: radiotherapy — Thoracic radiotherapy will begin no later than the start of the third chemotherapy cycle.
Radiation: Prophylactic Cranial Irradiation — PCI is recommended after the completion of chemoradiotherapy.
Drug: Consolidation Therapy with Toripalimab and Surufatinib — Patients achieving complete response (CR), partial response (PR), or stable disease (SD) following chemoradiotherapy will receive consolidation therapy. Toripalimab: 240 mg intravenously on day 1, every three weeks. Surufatinib: 200 mg orally on days 1-14, every three weeks.

SUMMARY:
Based on the preclinical rationale for combining surufatinib with immunotherapy, and the clinical efficacy observed with surufatinib in extensive-stage small cell lung cancer (ES-SCLC), the investigators hypothesize that incorporating surufatinib into the ADRIATIC regimen could further enhance survival in LS-SCLC. To evaluate this approach, the investigators plan to conduct a single-arm Phase II study to explore the safety and efficacy of concurrent chemoradiotherapy combined with toripalimab and surufatinib in treating LS-SCLC.

DETAILED DESCRIPTION:
This single-arm Phase II study aims to explore the safety and efficacy of concurrent chemoradiotherapy combined with toripalimab and surufatinib in treating LS-SCLC. In this single-arm, Phase II study, patients are planned to receive four cycles of etoposide combined with either cisplatin or carboplatin, along with toripalimab and surufatinib. During chemotherapy, patients will undergo concurrent radiotherapy. Following chemoradiotherapy, consolidation treatment with toripalimab and surufatinib will be administered. Prophylactic cranial irradiation (PCI) is recommended prior to the consolidation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent: An informed consent form, signed and dated, must be provided before any steps in the study are performed.
* Age: Males or females aged 18 to 75 years.
* Diagnosis: Histologically or cytologically confirmed small cell lung cancer (SCLC).
* Stage: Stage I-III (AJCC/UICC 8th edition TNM staging), where all lesions can be included in a single radical radiotherapy plan (i.e., limited-stage disease). Stage I-II must be inoperable.
* Life Expectancy: ≥12 weeks.
* Performance Status (PS): WHO PS score of 0 or 1.
* Postmenopausal women or those with a negative urine or serum pregnancy test (HCG sensitivity ≥25 IU/L or equivalent) within 7 days before starting study treatment.
* Female participants must not be breastfeeding.
* Women of childbearing potential (WOCBP) must agree to use contraception during study treatment and for 3 months after the last dose of study drug (i.e., 30 days for an ovulation cycle plus approximately 5 half-lives of the investigational drug).
* Male participants engaging in sexual activity with WOCBP must agree to use contraception during study treatment and for 5 months after the last dose of study drug (i.e., 90 days for sperm regeneration cycle plus approximately 5 half-lives of the investigational drug).
* Males with azoospermia do not need to follow contraception requirements.
* WOCBP who are not sexually active do not need to follow contraception requirements but must still undergo pregnancy testing as outlined.
* Organ and Bone Marrow Function:

Pulmonary Function: FEV1 ≥800 mL. Absolute neutrophil count ≥1.5 × 10⁹/L. Platelet count ≥100 × 10⁹/L. Hemoglobin ≥9.0 g/dL. Renal Function: Calculated creatinine clearance ≥50 mL/min using the Cockcroft-Gault formula.

Serum bilirubin ≤1.5 × upper limit of normal (ULN). AST and ALT ≤2.5 × ULN.

Exclusion Criteria:

* Participation in Another Clinical Trial: Simultaneous participation in another clinical trial, unless it is an observational (non-interventional) study.
* Mixed Histology: Histological subtype of mixed small cell and non-small cell lung cancer (SCLC).
* Extensive-Stage SCLC: Diagnosis of extensive-stage SCLC.
* Malignant Effusions: Pathologically confirmed malignant pleural effusion or pericardial effusion.
* Hemoptysis: Central cavitary SCLC with hemoptysis (hemoptysis volume >50 ml/day).
* Immunosuppressive Treatment: Use of immunosuppressive drugs within 28 days prior to the first dose of toripalimab. Physiological doses of intranasal corticosteroids and systemic corticosteroids ≤10 mg daily of prednisone (or equivalent) are exceptions. Steroids used to manage chemoradiotherapy-related toxicities are allowed.
* Previous Anti-PD-1/PD-L1 Therapy: Prior use of any anti-PD-1 or anti-PD-L1 antibodies.
* Major Surgery: Underwent major surgery (excluding vascular access) within 4 weeks before study entry.
* Autoimmune Disease History: History of autoimmune diseases within the last 2 years, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, or multiple sclerosis.
* Primary Immunodeficiency: History of primary immunodeficiency.
* Organ Transplant History: History of organ transplantation requiring immunosuppressive treatment.
* QT Interval Prolongation: QTc interval (corrected by Bazett's formula) >470 ms, calculated from three ECG measurements.
* Uncontrolled Comorbidities: Uncontrolled comorbid conditions, including but not limited to persistent or active infections, symptomatic congestive heart failure, poorly controlled hypertension, unstable angina, arrhythmias, active peptic ulcer disease or gastritis, active bleeding disorders, chronic hepatitis C, HIV infection, HBsAg-positive patients with DNA >500 IU/ml, or any psychiatric or social conditions that may interfere with study requirements or the patient's ability to provide informed consent.
* Tuberculosis History: Known history of tuberculosis.
* Live Vaccination: Received a live attenuated vaccine within 30 days prior to study initiation.
* Previous Primary Malignancy: History of another primary malignancy within 5 years prior to study entry, except for adequately treated basal or squamous cell carcinoma of the skin, in situ cervical cancer, ductal carcinoma in situ of the breast, or localized prostate cancer.
* Pregnancy and Breastfeeding: Pregnant or breastfeeding women, or men and women of reproductive potential who are not using effective contraception.
* Interference with Study Assessment: Any condition that may interfere with the evaluation of toripalimab's efficacy or safety.
* Investigator's Discretion: Any other condition that, in the opinion of the investigator, would make the patient unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2028-11-29 (Estimated); Study Completion 2028-11-29 (Estimated)

PRIMARY OUTCOMES:
Median progression-free survival (PFS) | 2 years
  The length of time from the start of treatment until disease progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Median overall survival (OS) | 2 years
  The time from the start of treatment to death from any cause.
Treatment-related adverse events | 1 year after treatment
  The assessment of treatment-related adverse events (AEs), including their type, severity, frequency, and impact on patients.
Patient-Reported Outcomes | 1 year after treatment
  Patient reported quality of life measured by European organization for Research and Treatment of Cancer (EORTC) Quality of Life Core 30 (QLQ-C30) and QLQ-LC13.

OTHER OUTCOMES:
Circulating Tumor DNA | 2 years
  The analysis of variations in ctDNA levels during and after treatment, and their correlation with patient outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Professor, Principal Investigator — Sun yat-sen universtiy cancer center
Locations (1):
- Sun yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Zhang Y, Huang Y, Yang Y, Zhao Y, Zhou T, Chen G, Zhao S, Zhou H, Ma Y, Hong S, Zhao H, Zhang L, Fang W. Surufatinib plus toripalimab combined with etoposide and cisplatin as first-line treatment in advanced small-cell lung cancer patients: a phase Ib/II trial. Signal Transduct Target Ther. 2024 Sep 27;9(1):255. doi: 10.1038/s41392-024-01974-2. PMID 39327433
- [Background] Li, X. et al. Enhanced anticancer efficacy via ROS-dependent ferroptosis: Synergy between surufatinib and cisplatin in small cell lung cancer. Cancer Res 84(6_Supplement), 2122 (2024)
- [Background] Zhou, J. et al. Preclinical evaluation of sulfatinib, a novel angio-immuno kinase inhibitor targeting VEGFR, FGFR-1 and CSF-1R kinases. AACR 77, abs 4187 (2017)
- [Background] David R. Spigel et al., ADRIATIC: Durvalumab (D) as consolidation treatment (tx) for patients (pts) with limited-stage small-cell lung cancer (LS-SCLC). JCO 42, LBA5-LBA5(2024).
- [Background] Senan S, Okamoto I, Lee GW, Chen Y, Niho S, Mak G, Yao W, Shire N, Jiang H, Cho BC. Design and Rationale for a Phase III, Randomized, Placebo-controlled Trial of Durvalumab With or Without Tremelimumab After Concurrent Chemoradiotherapy for Patients With Limited-stage Small-cell Lung Cancer: The ADRIATIC Study. Clin Lung Cancer. 2020 Mar;21(2):e84-e88. doi: 10.1016/j.cllc.2019.12.006. Epub 2019 Dec 28. PMID 31948903
- [Background] Takada M, Fukuoka M, Kawahara M, Sugiura T, Yokoyama A, Yokota S, Nishiwaki Y, Watanabe K, Noda K, Tamura T, Fukuda H, Saijo N. Phase III study of concurrent versus sequential thoracic radiotherapy in combination with cisplatin and etoposide for limited-stage small-cell lung cancer: results of the Japan Clinical Oncology Group Study 9104. J Clin Oncol. 2002 Jul 15;20(14):3054-60. doi: 10.1200/JCO.2002.12.071. PMID 12118018
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593